CLINICAL TRIAL: NCT05981313
Title: Evaluation of Viscoelastic Properties of Lower Extremity Muscles in Patients With Hemophilia
Brief Title: Viscoelastic Properties of Lower Extremity Muscles in Patients With Hemophilia
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hasan Kalyoncu University (Other)
Responsible Party: Principal Investigator, Tuğba GÖNEN, Assistant Professor, Hasan Kalyoncu University
Other Study IDs: 2023/52
Record Dates: First submitted 2023-07-16; First posted 2023-08-08 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-07

CONDITIONS: Hemophilia; Hemophilia A; Hemophilia B
Keywords: Hemophilia; Muscle tone; Stiffness; Elasticity
MeSH Terms: conditions — Hemophilia A; Hemophilia B

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hemophilia Group: The viscoelastic properties (tone, stiffness, elasticity) of the lower extremity muscles (Vastus Medialis Obliquus, Rectus Femoris, Vastus Lateralis, Biceps Femoris, Tibialis Anterior, Gastrocnemius) of hemophilia patients who meet the study criteria will be evaluated with the MyotonPro device (Myoton Ltd).
- Control Group: The viscoelastic properties (tone, stiffness, elasticity) of the lower extremity muscles (Vastus Medialis Obliquus, Rectus Femoris, Vastus Lateralis, Biceps Femoris, Tibialis Anterior, Gastrocnemius) of healthy children meeting the study criteria will be evaluated with the MyotonPro device (Myoton Ltd).

SUMMARY:
The aim of our study is to evaluate the viscoelastic properties of lower extremity muscles in patients with hemophilia A and hemophilia B secondarily to compare them with their healthy peers.

DETAILED DESCRIPTION:
Hemophilia is a rare inherited coagulation disorder that develops as a result of factor VIII (hemophilia A) or factor IX (hemophilia B) deficiency, and is a chronic group of diseases that mainly manifests with intra-articular (hemarthrosis) and intramuscular (hematoma) bleeding, affecting quality of life. The presence of easy ecchymosis formation in early childhood, especially intra-articular and intramuscular spontaneous bleeding, interventions and a history of bleeding that lasted longer than expected after trauma should suggest hemophilia. The severity of bleeding findings is directly related to the degree of deficiency of hemophilia A and B. Hemarthroses due to bleeding in the joint (80%) and hematomas due to intramuscular bleeding (20%) cause joint degeneration and muscle atrophy. The joint in which hemarthrosis is most common is the knee joint, however, bleeding into the lower extremity muscles seriously affects the activities of daily living and lower extremity functionality. For this reason, the researchers aimed to evaluate the viscoelastic properties of lower extremity muscles in hemophilia patients and, secondarily, to compare them with their healthy peers.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 4-17 years
* Those who have been diagnosed with Hemophilia A and Hemophilia B by a physician
* No history of acute bleeding
* Children who have family consent and volunteer to participate in the study

Exclusion Criteria:

* Those with a history of lower extremity surgery
* Those with neurological disease
* Those with a history of lower extremity hemarthrosis or hematoma in the last 1 month
* Patients with inhibitor positive

Ages: 4 Years to 17 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — Hemophilia A and B disease is an X-linked recessive disease. Therefore, girls become carriers and do not show muscle joint problems.
Study Population: Pediatric group hemophilia A and hemophilia B children living in Gaziantep constitute the study population.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2023-08-15 (Estimated); Primary Completion 2023-08-16 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Lower extremity moscle tone (Hz) | through of the study, average 6 months
  The tone (Hz) of lower extremity muscles (Vastus Medialis Obliquus, Rectus Femoris, Vastus Lateralis, Biceps Femoris, Tibialis Anterior, Gastrocnemius) will be evaluated with MyotonPro device (Myoton Ltd). Vastus Medialis Obliquus, Rectus Femoris, Vastus Lateralis and Tibialis Anterior muscle measurements will be made from the reference points determined in the supine relaxed position, while Biceps Femoris and Gastrocnemius measurements will be made in the prone position with the ankle in the neutral position. Participants will be allowed to rest on the table for 10 minutes before the measurements are taken. The viscoelastic measurement will be repeated three times by determining the reference points (cm) of the relevant muscles and the averages will be recorded. Only measurements with a coefficient of variation less than 3% will be taken into account, otherwise the measurements will be repeated.
Lower extremity stiffness (N/m) | through of the study, average 6 months
  The stiffness (N/m) of lower extremity muscles (Vastus Medialis Obliquus, Rectus Femoris, Vastus Lateralis, Biceps Femoris, Tibialis Anterior, Gastrocnemius) will be evaluated with MyotonPro device (Myoton Ltd). Vastus Medialis Obliquus, Rectus Femoris, Vastus Lateralis and Tibialis Anterior muscle measurements will be made from the reference points determined in the supine relaxed position, while Biceps Femoris and Gastrocnemius measurements will be made in the prone position with the ankle in the neutral position. Participants will be allowed to rest on the table for 10 minutes before the measurements are taken. The viscoelastic measurement will be repeated three times by determining the reference points (cm) of the respective muscles and the averages will be recorded. Only measurements with a coefficient of variation less than 3% will be taken into account, otherwise the measurements will be repeated.
Lower extremity elasticity (log) | through of the study, average 6 months
  The elasticity (log) of lower extremity muscles (Vastus Medialis Obliquus, Rectus Femoris, Vastus Lateralis, Biceps Femoris, Tibialis Anterior, Gastrocnemius) will be evaluated with MyotonPro device (Myoton Ltd). Vastus Medialis Obliquus, Rectus Femoris, Vastus Lateralis and Tibialis Anterior muscle measurements will be made from the reference points determined in the supine relaxed position, while Biceps Femoris and Gastrocnemius measurements will be made in the prone position with the ankle in the neutral position. Participants will be allowed to rest on the table for 10 minutes before the measurements are taken. The viscoelastic measurement will be repeated three times by determining the reference points (cm) of the respective muscles and the averages will be recorded. Only measurements with a coefficient of variation less than 3% will be taken into account, otherwise the measurements will be repeated.

CONTACTS AND LOCATIONS:
Locations (1):
- Hasan Kalyoncu University, Gaziantep, Şahinbey, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Srivastava A, Santagostino E, Dougall A, Kitchen S, Sutherland M, Pipe SW, Carcao M, Mahlangu J, Ragni MV, Windyga J, Llinas A, Goddard NJ, Mohan R, Poonnoose PM, Feldman BM, Lewis SZ, van den Berg HM, Pierce GF; WFH Guidelines for the Management of Hemophilia panelists and co-authors. WFH Guidelines for the Management of Hemophilia, 3rd edition. Haemophilia. 2020 Aug;26 Suppl 6:1-158. doi: 10.1111/hae.14046. Epub 2020 Aug 3. No abstract available. PMID 32744769
- [Background] Schafer GS, Valderramas S, Gomes AR, Budib MB, Wolff AL, Ramos AA. Physical exercise, pain and musculoskeletal function in patients with haemophilia: a systematic review. Haemophilia. 2016 May;22(3):e119-29. doi: 10.1111/hae.12909. Epub 2016 Apr 14. PMID 27075748
- [Background] De la Corte-Rodriguez H, Rodriguez-Merchan EC. The role of physical medicine and rehabilitation in haemophiliac patients. Blood Coagul Fibrinolysis. 2013 Jan;24(1):1-9. doi: 10.1097/MBC.0b013e32835a72f3. PMID 23103725
- [Background] Usgu S, Ramazanoglu E, Yakut Y. The Relation of Body Mass Index to Muscular Viscoelastic Properties in Normal and Overweight Individuals. Medicina (Kaunas). 2021 Sep 26;57(10):1022. doi: 10.3390/medicina57101022. PMID 34684059